CLINICAL TRIAL: NCT05714189
Title: The Effect of Dietary Interventions, or no Intervention, on Pain and Quality of Life in Women Diagnosed With Endometriosis
Acronym: Dieetstudie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof. Velja Mijatovic, Professor Doctor, Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: W20_534 # 20.593
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — FODMAP Diet

STUDY DESIGN:
Intervention Model Description: Women could chose to adhere to a diet or the control group. there was no cross-over.
Masking Description: Women were able to choose themselves whether to adhere to a diet, and to which diet, or to adhere to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group: adherence to Low FODMAP diet (Other): Women could choose to adhere to the low FODMAP diet, over a period of six months. In the first three months, they received extensive guidance by a dietician in training, in addition to supportive materials such as the Monash app, recipes and grocery lists, in the hope of optimal adherence to the diet. After three months, women were asked to continue the diet independently. In addition, women were asked to complete three questionnaires, one every two months. The questionnaires contained the EHP-30, the GIQLI, and self composed questions on their demographics in the first questionnaire, and their strictness of adherence in the second and third questionnaire. The third questionnaire also contained questions on their satisfaction with the dietary guidance and the dietician in training.
  Interventions: Other: Low FODMAP diet
- Intervention group: adherence to endometriosis diet (Other): Women could choose to adhere to the endometriosis diet, over a period of six months. In the first three months, they received extensive guidance by a dietician in training, in addition to supportive materials such as the Monash app, recipes and grocery lists, in the hope of optimal adherence to the diet. After three months, women were asked to continue the diet independently. In addition, women were asked to complete three questionnaires, one every two months. The questionnaires contained the EHP-30, the GIQLI, and self composed questions on their demographics in the first questionnaire, and their strictness of adherence in the second and third questionnaire. The third questionnaire also contained questions on their satisfaction with the dietary guidance and the dietician in training.
  Interventions: Other: Endometriosis diet
- Control group: no diet adherence (No Intervention): Women were asked to complete three questionnaires, once every two months. These contained the EHP-30 and GIQLI. The first questionnaire contained questions on their demographics, and whether they applied a diet before.

INTERVENTIONS:
Other: Low FODMAP diet — The Low FODMAP diet is an avoidance diet and consist of three phases. In the first phase, all nutrients high in FODMAPs (high-FODMAPS) are eliminated from the daily diet over a period of 2 to 6 weeks to calm down the bowel. The second phase consists of the addition of FODMAP challenges. During this phase the patient continues the Low FODMAP diet, but will reintroduce one high-FODMAP nutrient once every three days to see whether exposure to this high-FODMAP causes IBS symptoms. When this is not the case, the patient can continue eating this high-FODMAP group in their daily diet. In the third and final phase, the diet is fully personalized. This personalization is based on whether the patient tolerated the high-FODMAP nutrient or not during the FODMAP challenges. Only when the high-FODMAP nutrient is not tolerated, it is advised to permanently remove it from the daily diet.
  Arms: Intervention group: adherence to Low FODMAP diet
Other: Endometriosis diet — The endometriosis diet The endometriosis diet is a patient experience based, avoidance diet developed by women diagnosed with endometriosis. Therefore no specific recommendations exist regarding the application of the endometriosis diet. With the endometriosis diet, women avoid nutrients they noticed provoked or aggravated their endometriosis-related symptoms such as red meat, coffee, sugar, lactose and soy.
  Arms: Intervention group: adherence to endometriosis diet

SUMMARY:
This prospective pilot study was performed to explore the influence of a dietary intervention, the Low FODMAP diet or endometriosis diet, on endometriosis-related pain and Quality of Life (QoL). Participants could choose between adherence to a diet; the Low FODMAP diet or endometriosis diet, or to contribute to the control group and not adhere to a diet.

DETAILED DESCRIPTION:
This prospective pilot study was performed to explore the influence of a dietary intervention, the Low FODMAP diet or endometriosis diet, on endometriosis-related pain and Quality of Life (QoL). Participants could choose between adherence to a diet; the Low FODMAP diet or endometriosis diet, or to contribute to the control group and not adhere to a diet. Women choosing to adhere to a diet were extensively guided by a dietician in training. In addition, both groups are asked to complete three questionnaires over a period of six months; once every two months.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with endometriosis, either through radiologic imaging (transvaginal ultrasound and/or MRI) or laparoscopy
* A reported pain score of ≥ 3 (Visual Analogue Score (VAS), scale 0-10cm) in one or more of the following symptoms: dysmenorrhea, deep dyspareunia and chronic pelvic pain

Exclusion Criteria:

* about to undergo an operation within six months
* Undergone an operation in the past six weeks
* a switch in hormonal therapy within six weeks
* Women that were pregnant or breastfeeding
* women diagnosed with a malignancy
* An additional diagnosis with Coeliac Disease (CD) and/or lactose intolerance.
* Not sufficient in the Dutch or English language.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women diagnosed with endometriosis
Enrollment: 62 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
pain scores | 6 months
  The primary outcome focused on pain scores (in VAS, scale 0-10cm) of the endometriosis-related symptoms dysmenorrhea, deep dyspareunia, chronic pelvic pain, dysuria, dyschezia, tiredness and bloating. Pain scores will be measured on a scale between 0 and 10, where 0 represents no pain at all and 10 the worst pain possible.

SECONDARY OUTCOMES:
Quality of Life (QoL) | 6 months
  Secondary outcome focused on QoL, expressed using the EHP-30 questionnaire. Using the EHP-30, a score between 0 and 100 can be measured for 11 different QoL domains. For every domain, a score of 0 represents best health status through to a score of 100 which represents worst health status.
Gastro-Intestinal Health | 6 months
  Secondary outcome focused on gastro-intestinal health, expressed using the GIQLI questionnaire. With the GIQLI, a score between 0 and 144 can be calculated where 0 represents worst possible gastro-intestinal health and 144 best possible gastro-intestinal health.
Adhesion to dietary intervention | 6 months
  with every follow-up visit, women were asked on their dietary adhesion. they were asked how often they made an exception, with what meal (snack/main meal) and what strictness score they gave themselves. Women could score their strictness between 0 and 10 where 0 represented worst possible strictness and 10 best possible strictness

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No